CLINICAL TRIAL: NCT03157882
Title: Pediatric Pain Assessment in the Emergency Department
Status: Terminated | Type: Observational
Why Stopped: loss of funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 09-16-31E
Record Dates: First submitted 2017-05-11; First posted 2017-05-17 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2019-08

CONDITIONS: Pain; Acute Pain
Keywords: pediatric; children; Faces Pain Scale Revised; Wong Baker FACES; pain scales; BRIGANCE
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Population: Pediatric patients presenting to the emergency department with acute painful conditions (please see inclusion and exclusion criteria)

SUMMARY:
To examine pediatric pain assessment in the Emergency Department

DETAILED DESCRIPTION:
Phase 1 is a qualitative assessment of how pain is currently evaluated in the pediatric Emergency Department (ED). Initial triage encounters will be observed and audio recorded. In addition to determining how often the Wong Baker FACES Pain Rating Scale (WBF) is administered with the intended script, the investigators will determine if there are common variations from the recommended script. The investigators will also evaluate how often a caregiver's perception of the child's pain is considered when completing the WBF.

Phase 2 is a quantitative assessment to determine if neurocognitive development impacts the responsivity of the WBF and the Faces Pain Scale - Revised (FPS-R) as well as the cognitive age equivalent required to use these scales accurately. Patients presenting with acute pain will report their level of pain before and after analgesic intervention using both the WBF and the FPS-R. They will also subjectively report their change in pain following analgesic intervention. Once the patient's pain has improved, he/she will complete the BRIGANCE Early Childhood Screens III to determine his/her cognitive age equivalent. He/she will also complete a series of tasks aimed to assess ability to successfully use the WBF and FPS-R (matching, grouping, classification, and seriation skills). The results of the child's self-report of pain will also be compared to the caregiver's estimate of the child's pain.

ELIGIBILITY:
Inclusion Criteria:

* verbal patients
* pain score ≥ 6/10
* caregiver speaks English or Spanish

Exclusion Criteria:

* altered mental status
* history of traumatic brain injury (TBI)
* history of developmental delay
* history of Autism
* history of chronic pain, defined as persistent or recurrent pain in children with chronic health conditions
* non-verbal patients

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients presenting to the emergency department with complaint of pain
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-08-13 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Qualitative Assessment (Phase 1 - Primary Aim) | One day
  Adherence to a validated script for pain scale administration (dichotomous value - yes/no)
Wong-Baker FACES ® Pain Rating Scale (WBF) | One day
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Change in pain scale response before and after analgesic intervention that correlates with a subjective description of change in pain (better or worse).
Faces Pain Scale - Revised (FPS-R) | One day
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Change in pain scale response before and after analgesic intervention that correlates with a subjective description of change in pain (better or worse).

SECONDARY OUTCOMES:
Convergent reliability between WBF and FPS-R (Phase 2 Secondary Aim #1) | One day
  Convergent reliability between WBF and FPS-R - determined by pre and post analgesia reports of pain using the FPS-R and WBF by the patient. Both scales show a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable".
Pre and Post Analgesia Pain Scores Using WBF and FPS-R as Reported by Patients and Caregivers | One day
  Inter-rater reliability between children and caregivers when using WBF and FPS-R, determined by pre and post analgesia reports of pain using the FPS-R and WBF by both the patient and caregiver. Both scales show a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Simone L Lawson, MD, Principal Investigator — Wake Forest University Health Sciences; Melanie Hogg, Study Director — Wake Forest University Health Sciences
Locations (1):
- Simone Lorraine Lawson, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT03157882/Prot_SAP_000.pdf